CLINICAL TRIAL: NCT00386087
Title: A Phase II Study of Oral Enzastaurin in Patients With Metastatic Breast Cancer Previously Treated With an Anthracycline and a Taxane-Containing Regimen
Brief Title: Enzastaurin For Breast Cancer Patients Who Previously Received an Anthracycline and a Taxane Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10517; H6Q-MC-S015
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-04

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Drug: Enzastaurin Hydrochloride

SUMMARY:
The purpose of this study is to determine the effectiveness of enzastaurin in the treatment of patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of metastatic breast cancer or recurrent breast cancer where surgery can not be done for curative intent
* Have received prior therapy with an anthracycline (class of drugs) and a taxane (class of drugs).
* Tumors must not be positive for HER2, but if positive, the treatment plan should not include further treatment with the drug Herceptin.
* Disease that can be definitely measured on Cat Scans or other radiological tests.
* May have received high dose chemotherapy for autologous stem cell support greater than or equal to 6 months of starting this study.

Exclusion Criteria:

* More than 2 chemotherapy regimens for metastatic or locally recurrent disease.
* Have brain cancer from breast cancer
* Pregnant or breastfeeding
* Have an inability to swallow tablets
* Within 6 months have had a serious heart condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2006-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To determine the effects of enzastaurin in the treatment of patients with breast cancer by measuring its ability to reduce the size of the tumor or prevent further increases in tumor size.

SECONDARY OUTCOMES:
To evaluate the length of time that enzastaurin is able to effect control of the disease.
To evaluate the side effects of enzastaurin in patients with breast cancer
To determine whether changes in laboratory tests of patients treated with enzastaurin is associated with the response of their tumors to the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time(UTC/GMT - 5 Hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newark, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Bend, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts

REFERENCES:
- See also: Hoosier Oncology Group — http://www.hoosieroncologygroup.org
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com